CLINICAL TRIAL: NCT03386045
Title: Optimal Prostate Fractionation Study
Brief Title: Optimal Prostate Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMAL
Record Dates: First submitted 2017-12-11; First posted 2017-12-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal SBRT (Active Comparator): Participants in this group will be randomised to either SBRT ( 36 to 45 GY in 5 fractions) or standard radiotherapy (60 Gy in 20 fractions). The allocation is 2 to 1. This means that two thirds of the participants on the trial will get the SBRT (5 treatments) and one third will get the standard fractions.
  Interventions: Radiation: Optimal SBRT
- Optimal Booster (Active Comparator): Participants in this group will be randomised to either standard radiotherapy plus SBRT (45 Gy in 20 fractions plus 20-30 Gy in 2 fractions-Booster) or standard radiotherapy (60 Gy in 20 fractions). The allocation is 2 to 1. This means that two thirds of the participants on the trial will get the Booster arm and one third will get the standard fractions.
  Interventions: Radiation: Optimal Booster

INTERVENTIONS:
Radiation: Optimal SBRT — Two thirds of the participants in this group will get the SBRT (5 treatments) and one third will get standard treatment (60 Gy in 20 treatments)
  Arms: Optimal SBRT
Radiation: Optimal Booster — Two thirds of the participants in this group will get the two high precision radiotherapy plus 20 doses of standard external beam radiotherapy (ie the "Booster approach|") and one third will get the standard treatment (60 Gy in 20 treatments)
  Arms: Optimal Booster

SUMMARY:
To compare the toxicity, rate of local control, biochemical failure rate and quality of life of three different radiotherapy techniques (moderate hypofractionation, stereotactic body radiotherapy (SBRT) and standard radiotherapy plus 2 fractions of SBRT (BOOSTER)

DETAILED DESCRIPTION:
Participants must have histologically proven prostate adenocarcinoma, good performance status and suitable for high dose radiotherapy. There are two groups of participants:

Group 1: eligible participants will be randomised to have either moderate hypofractionation or standard radiotherapy plus SBRT (BOOSTER). Participants in this group must be able to have MRI, prostate fiducial markers (gold markers)and hydrogel insertion. Fiducial markers will be used to locate the prostate accurately during radiation treatment. Hydrogel is a temporary gel being injected into the space between the prostate and rectum to reduce the dose of radiation received by the rectum to minimise side effects from the treatment.

Group 2: eligible participants will be randomised to have either moderate hypofractionation or SBRT.

Participants will be reviewed for side effects. A Safety Committee will be formed containing multi-disciplinary team members. All serious adverse will be reported to the principal investigator and Human Research Ethics Committee within 24 hours.

ELIGIBILITY:
Inclusion criteria

* Histologically proven prostate adenocarcinoma
* PSA obtained within three months prior to enrolment
* ECOG performance status 0 to 2
* Ability to understand and the willingness to sign a written consent
* Suitable for high dose irradiation to the prostate

To be eligible for the arm containing Stereotactic Booster alone approach patient must have the following

* No contraindication to MRI such as pacemaker and severe claustrophobia
* Patient must be able to have fiducial markers placed in the prostate
* Patient must be able to have hydrogel insertion at the same time as fiducial markers
* Must have IPSS less than 15

Exclusion criteria

* Previous pelvic radiotherapy
* Prior total prostatectomy
* Unwilling or unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
local control | 12 months post radiotherapy
  the rate of local control as determined on PSMA scanning

SECONDARY OUTCOMES:
Biological failure rate | 3 year and 5 year
  The rate of biochemical failure defined as Nadir+2.0 biochemical failure defined as Nadir+2.0
late toxicity | more than three months after treatment completion.
  Late Gastrointestinal and Genitourinary Toxicity (modified RTOG scale)
Markerless tracking technology | During radiotherapy treatment
  Markerless tracking algorithms will be assessed for accuracy against marker-based localisation by masking the markers and directly comparing the determined trajectories
Accuracy of the various intrafraction guidance methods | During radiotherapy treatment
  Accuracy of various intrafraction guidance methods will be determined against triangulation of kilovoltage (kV) and Megavoltage (MV) projections

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kneebone, MBBS, Principal Investigator — Northern Sydney Local Health District
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
aim to present study data in conferences and medical journals
Time Frame: end of trial after analysis